CLINICAL TRIAL: NCT01054144
Title: Phase II Study of Response Adapted Therapy Using Single Agent Lenalidomide in Older Adults With Newly Diagnosed, Standard Risk Multiple Myeloma
Brief Title: Study of Single Agent Lenalidomide in Older Adults With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16018; 108562 (Other: USF IRB); RV-MM-PI-0454 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed Standard Risk Multiple Myeloma; Senior Adults
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Prednisone; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Response Adapted Therapy (Experimental): Lenalidomide, prednisone and dexamethasone as outlined in Intervention Descriptions.
  Interventions: Drug: Lenalidomide; Drug: Prednisone; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — * Starting Dose: 25 mg by mouth (PO) days 1-21 of a 28 days cycle;
  * Dose Level -1: 15 mg PO days 1-21 of a 28 days cycle;
  * Dose Level -2: 10 mg PO days 1-21 of a 28 days cycle;
  * Dose Level -3: 5 mg PO days 1-21 of a 28 days cycle;
  * Dose Level -4: Discontinue
  Other Names: Revlimid®
Drug: Prednisone — * Starting Dose: 100 mg PO days 1-5 every 28 days;
  * Dose level -1: 50 mg PO days 1-5 of a 28 day cycle;
  * Dose level -2: 25 mg PO days 1-5 of a 28 day cycle;
  * Dose level -3: Discontinue
Drug: Dexamethasone — * Starting Dose: 40 mg daily on days 1 - 4 every 28 days;
  * Dose level -1: 20 mg daily on days 1 - 4 every 28 days;
  * Dose level -1a: 40 mg daily on days 1, 2, and 3 followed by 20 mg on day 4 followed by 12 mg on day 5 followed by 8 mg on day 6;
  * Dose level -2: 10 mg daily on days 1 - 4 every 28 days;
  * Dose level -3: Discontinue
  Other Names: Decadron

SUMMARY:
The purpose of this research is to estimate the effectiveness of a response adapted approach with the use of the drug, lenalidomide in the treatment of older adults with newly diagnosed standard risk multiple myeloma. This means that participants will be given the study drug, lenalidomide but depending on how they respond to this drug they may also be given dexamethasone and/or prednisone to help with their treatment.

DETAILED DESCRIPTION:
Summary: Patients will be started on the study drug, lenalidomide on Day 1, Cycle 1. Lenalidomide is a capsule that is to be taken orally (by mouth). If the patient's disease progresses after 2 cycles of therapy, a low dose of dexamethasone will be added. If the patient's disease is stable after 2 cycles of therapy, the use of an alternate corticosteroid (prednisone) will be added to the lenalidomide therapy they are receiving. Dexamethasone and prednisone are in tablet form and will be taken orally (by mouth). However, if the patient has a minimal response after an additional 2 cycles of lenalidomide therapy, the therapy will be continued until their disease progresses. See the intervention descriptions for further details.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Age ≥65 years or not eligible for high dose therapy and autologous stem cell transplant
* Able to adhere to study visit schedule and other protocol requirements
* Diagnosed with multiple myeloma and considered to have active disease. Patients must not have received an active chemotherapy regimen or Dexamethasone. Patients may have received palliative radiotherapy at least 2 weeks prior to the study start.
* Measurable myeloma paraprotein levels in serum (≥ 0.5 g/dL), urine (≥ 0.2 g excreted in a 24-hour urine collection sample) or by serum free light chains (involved free light chain greater than 100mg/L)
* Eastern Cooperative Group (ECOG) Performance Status of 0 or 1
* Serum bilirubin levels ≤1.5 times the upper limit of the normal (ULN) range for the laboratory
* Serum aspartate transaminase (AST) or serum alanine transaminase (ALT) levels ≤2 x ULN
* Adequate bone marrow function: Absolute neutrophil count ≥ 1,000 cells/mm³ (1.0 x 10^9/L); Platelets ≥ 100,000 /mm³
* Hemoglobin > 8 g/dL
* Adequate renal function: Calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula
* Low risk myeloma is defined as the absence of the following adverse features[21]: t(4;14) by FISH or metaphase cytogenetics; t(14,16) or t(14;20) by FISH or metaphase cytogenetics; Deletion 17q13 by FISH; Deletion 13 by metaphase analysis; Aneuploidy by metaphase analysis; Β2 microglobulin > 5.5.
* Able to tolerate one of the following thromboprophylactic strategies: aspirin, low molecular weight heparin or warfarin (coumadin)
* Must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-international units per milliliter (mIU/mL) within 10 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy.

Exclusion Criteria:

* Ongoing severe infection requiring intravenous antibiotic treatment
* Life expectancy of less than 3 months
* Performance status of 2, 3 or 4
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer from which the patient has been disease-free for at least 2 years
* Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia
* Uncontrolled medical problems such as diabetes mellitus, congestive heart failure, coronary artery disease, hypertension, unstable angina, arrhythmias), pulmonary, hepatic and renal diseases unless renal insufficiency is felt to be secondary to multiple myeloma.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or lactating
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Known hypersensitivity to thalidomide
* Use of any other experimental drug or therapy within 28 days of baseline.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-01-14 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachid Baz, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Response Adapted Therapy: Lenalidomide, prednisone and dexamethasone as outlined in Intervention Descriptions.
  Lenalidomide: - Starting Dose: 25 mg by mouth (PO) days 1-21 of a 28 days cycle;
  * Dose Level -1: 15 mg PO days 1-21 of a 28 days cycle;
  * Dose Level -2: 10 mg PO days 1-21 of a 28 days cycle;
  * Dose Level -3: 5 mg PO days 1-21 of a 28 days cycle;
  * Dose Level -4: Discontinue
  Prednisone: - Starting Dose: 100 mg PO days 1-5 every 28 days;
  * Dose level -1: 50 mg PO days 1-5 of a 28 day cycle;
  * Dose level -2: 25 mg PO days 1-5 of a 28 day cycle;
  * Dose level -3: Discontinue
  Dexamethasone: - Starting Dose: 40 mg daily on days 1 - 4 every 28 days;
  * Dose level -1: 20 mg daily on days 1 - 4 every 28 days;
  * Dose level -1a: 40 mg daily on days 1, 2, and 3 followed by 20 mg on day 4 followed by 12 mg on day 5 followed by 8 mg on day 6;
  * Dose level -2: 10 mg daily on days 1 - 4 every 28 days;
  * Dose level -3: Discontinue
Period: Overall Study
Arm/Group | Response Adapted Therapy
Started | 27
Completed | 25
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Response Adapted Therapy
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Combined Therapy - Median Progression Free Survival
Description: Progression free survival (PFS) of older adults with mildly symptomatic multiple myeloma treated on this response adapted approach (i.e. time from start of lenalidomide to failure of lenalidomide and low dose dexamethasone)
Time Frame: up to 36 months
Population: Number of participants who received response adaptive therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Response Adapted Therapy
Number analyzed (Participants) | 9
months | 36 [29.7 to NA] — Not reached

2. Secondary Outcome: Response Rate
Description: Response rate in older adults with mildly symptomatic multiple myeloma to single agent lenalidomide, lenalidomide prednisone and lenalidomide low dose dexamethasone in patients with suboptimal responses to lenalidomide monotherapy. The study used the uniform response assessment of the International Myeloma Working Group with the addition of MR (minimal response) (Durie et al, 2006; Kumar et al, 2016). MR was defined as a 25-49% decrease in serum M spike, and a 50-89% improvement in urine M spike. For patients without a measurable serum or urine M spike, a 25-49% decrease in the difference between the involved and uninvolved free light chains was required. The response in this trial is defined as complete remission (CR), stringent complete remission (SRC), very good partial remission (VGPR) and partial remission (PR) and minimal response (MR).
Time Frame: Every 8 weeks up to 12 months
Population: 1 participant could not be evaluated for response.
Measure: Count of Participants; unit: Participants
Groups:
- Single Agent Lenalidomide: Participants treated with single agent lenalidomide
Arm/Group | Response Adapted Therapy | Single Agent Lenalidomide
Number analyzed (Participants) | 9 | 26
Participants
  Complete Response & Stringent Complete Response | 1 | 4
  Very Good Partial Response (VGPR) | 1 | 3
  Partial Response (PR) | 2 | 12
  Minimal Response (MR) | 5 | 4
  Stable Disease | 0 | 3
  Overall Response >/= PR | 4 | 19

3. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants with serious adverse events
Time Frame: Day 1 through Off Study Date, an average of 48 months
Measure: Number; unit: participants
Arm/Group | Response Adapted Therapy
Number analyzed (Participants) | 27
participants | 20

4. Secondary Outcome: Single Agent - Median Progressive Free Survival (PFS)
Description: The progression free survival of patients treated with single agent lenalidomide
Time Frame: First measure at 8 weeks
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Single Agent: Participants who were treated with single agent lenalidomide only
Arm/Group | Single Agent
Number analyzed (Participants) | 18
months | 29 [25.7 to 73.5]

5. Secondary Outcome: Number of Participants With 1 Year Overall Survival (OS)
Description: The 1 year overall survival of older adults with mildly symptomatic multiple myeloma treated on this response adapted approach
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | Response Adapted Therapy
Number analyzed (Participants) | 27
participants | 27

ADVERSE EVENTS:
Time Frame: Adverse Events collected from consent through off treatment date, an average of 24 months. Serious Adverse events collected from consent to off-study date, an average of 48 months
Groups:
- All Participants: All participants treated with Lenalidomide, prednisone and lenalidomide, prednisone and dexamethasone as outlined in Intervention Descriptions.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 2/27
Serious Adverse Events (participants affected / at risk) | 20/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=27)
General Cardiac Disorders - Other (Cardiac disorders) | 3 (4)
Hypertension (Cardiac disorders) | 1 (2)
Hypotension (Cardiac disorders) | 2 (2)
Coagulation (General disorders) | 1 (1)
General disorders - Other (General disorders) | 1 (1)
Fever (General disorders) | 1 (2) — Fever in the absence of neutropenia where neutropenia is defined as ANC <1.0 x 10e9/L
Death (General disorders) | 1 (1) — Death not associated with CTCAE term - Sudden death
Wound complication (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders, other (Gastrointestinal disorders) | 1 (1)
Colon Obstruction (Gastrointestinal disorders) | 1 (1)
Hemorrhage, CNS (Vascular disorders) | 1 (1)
Hemorrhage, Stomach (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Colitis, Infectious (e.g. Clostridium difficile) (Infections and infestations) | 2 (2)
Febrile neutropenia (Infections and infestations) | 3 (3)
Infection -Blood (Infections and infestations) | 2 (2)
Infection - Lung (Infections and infestations) | 3 (3)
Infection - Other (Infections and infestations) | 1 (2)
Cellulitis (Infections and infestations) | 3 (3)
Infection - Bladder (Infections and infestations) | 1 (1)
Hypercalcemia (Investigations) | 1 (1)
Hyperglycemia (Investigations) | 1 (1)
Investigations -Other (Investigations) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Cerebrovascular ischemia (Vascular disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Mental status (Psychiatric disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Chest wall pain (General disorders) | 1 (1)
Limb pain (General disorders) | 2 (2)
Pain -Other (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vascular -Other (Vascular disorders) | 1 (3)
Non-myocardial vascular arterial ischemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=27)
Constipation (Gastrointestinal disorders) | 24 (46)
Diarrhea (Gastrointestinal disorders) | 23 (66)
Nausea (Gastrointestinal disorders) | 17 (37)
Anorexia (Metabolism and nutrition disorders) | 12 (27)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 12 (13)
Vomiting (Gastrointestinal disorders) | 11 (14)
Dehydration (Gastrointestinal disorders) | 9 (12)
Heartburn/dyspepsia (Gastrointestinal disorders) | 7 (9)
Distension/bloating, Abdominal (Gastrointestinal disorders) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Mucositis/stomatitis - oral cavity (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Obstruction, GI - Colon (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 23 (63)
Insomnia (General disorders) | 13 (20)
Fever (in absence of neutropenia) (General disorders) | 10 (25)
Weight loss (Metabolism and nutrition disorders) | 8 (11)
Rigors/chills (General disorders) | 5 (7)
Diaphoresis (General disorders) | 4 (4)
Weight gain (Metabolism and nutrition disorders) | 4 (4)
Constitutional symptoms - Other (General disorders) | 3 (3)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 25 (265)
Leukopenia (Blood and lymphatic system disorders) | 22 (264)
Low platelet count (Blood and lymphatic system disorders) | 20 (78)
Hemoglobin, low (Blood and lymphatic system disorders) | 16 (75)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Skin and subcutaneous tissue disorders -Other (Skin and subcutaneous tissue disorders) | 14 (27)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 14 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (18)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 10 (18)
Rash, erythema multiforme (Skin and subcutaneous tissue disorders) | 10 (16)
Brusing (Skin and subcutaneous tissue disorders) | 9 (13)
Flushing (Vascular disorders) | 5 (8)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (3)
Rash, acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Dermatitis associated with chemoradiation
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (General disorders) | 21 (45)
Pain - extremity/limb (General disorders) | 16 (29)
Headache (General disorders) | 16 (26)
Abdominal Pain NOS (Gastrointestinal disorders) | 12 (18)
Joint pain (General disorders) | 10 (12)
Chest wall pain (General disorders) | 6 (7)
Chest/thorax pain (General disorders) | 5 (7)
Neck pain (General disorders) | 5 (7)
Pain-throat/pharynx/larynx (General disorders) | 5 (6)
Pain - stomach (General disorders) | 4 (4)
Pain - muscle (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain - NOS (General disorders) | 3 (3)
Bone pain (General disorders) | 2 (3)
Pain - lymph node (General disorders) | 2 (2)
Pain - oral, gum (General disorders) | 2 (4)
Breast pain (General disorders) | 1 (1)
Buttock pain (General disorders) | 1 (1)
Pain - dental (General disorders) | 1 (1)
Pain - external ear (Ear and labyrinth disorders) | 1 (1)
Pain - eye (Eye disorders) | 1 (2)
Pain - face (General disorders) | 1 (1)
Gallbladder pain (Gastrointestinal disorders) | 1 (1)
Oral cavity pain (General disorders) | 1 (1)
Pelvic pain (General disorders) | 1 (1)
Sinus pain (General disorders) | 1 (1)
Pain - testicle (General disorders) | 1 (1)
Neuropathy, sensory (Nervous system disorders) | 19 (38)
Dizziness (Nervous system disorders) | 15 (29)
Nervous system disorders -Other (Nervous system disorders) | 9 (15)
Tremor (Nervous system disorders) | 8 (16)
Depression (Psychiatric disorders) | 6 (9)
Neuropathy, motor (Nervous system disorders) | 5 (6)
Agitation/Iritability (Psychiatric disorders) | 6 (8)
Anxiety (Psychiatric disorders) | 3 (6)
Confusion (Nervous system disorders) | 2 (3)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Neuropathy, cranial (Nervous system disorders) | 1 (1) — CN VIII hearing and balance
Personality/Behavior changes (Psychiatric disorders) | 1 (1)
Speech impairment (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Cough (Reproductive system and breast disorders) | 16 (28)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (25)
Respirator, thoracic and mediastrinal disorders -Other (Respiratory, thoracic and mediastinal disorders) | 9 (14)
Loss or alteration of voice (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paranasal/sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstruction of airway (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema - limb (General disorders) | 21 (52)
Edema -head and neck (General disorders) | 3 (4)
Edema - trunk (General disorders) | 1 (1)
Musculoskeletal and connective tissue disorders - Other (Musculoskeletal and connective tissue disorders) | 12 (19)
Muscle weakess, generalized (Musculoskeletal and connective tissue disorders) | 11 (12)
Muscle weakness, extraocular (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness, lower extremities (Musculoskeletal and connective tissue disorders) | 3 (3)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (3)
Gait changes (General disorders) | 5 (8)
Muscle weakness, trunk (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 6 (7)
Cellulitis (Infections and infestations) | 9 (11)
Infection -Other (Infections and infestations) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 4 (4)
Bronchus infection (Infections and infestations) | 3 (3)
Eye infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Sinus infection (Infections and infestations) | 3 (3)
Upper airway infection (Infections and infestations) | 1 (1)
Conjunctiva infection (Infections and infestations) | 2 (2)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Gingivitus (General disorders) | 2 (2)
Nail infection (Infections and infestations) | 1 (1)
wound infection (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Colon infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Hyperglycemia (Investigations) | 9 (13)
Creatinine (Investigations) | 7 (14)
Hyperkalemia (Investigations) | 7 (8)
ALT, SGPT high (Investigations) | 4 (6)
Hyperbilirubinemia (Investigations) | 4 (9)
Hypoalbuminemia (Investigations) | 3 (4)
Alkaline phosphatase (Investigations) | 3 (3)
Hypokalemia (Investigations) | 3 (5)
Investigations - Other (Investigations) | 11 (12)
Hypercalcemia (Investigations) | 2 (3)
Hypocalcemia (Investigations) | 2 (5)
Hypoglycemia (Investigations) | 2 (2)
AST, SGOT (Investigations) | 1 (1)
Hypomagnesemia (Investigations) | 1 (1)
Hypernatremia (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT01054144/Prot_SAP_000.pdf